CLINICAL TRIAL: NCT04238780
Title: Ultrasound Guided Erector Spinae Plane Block Reduces Postoperative Pain Following Laparoscopic Colorectal Operation: A Randomized Controlled Study
Brief Title: Erector Spinae Plane Block Reduces Postoperative Pain Following Laparoscopic Colorectal Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Jung Ju Choi, assistance professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESPlapaAR
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP( Erector Spinae Plane Block) (Active Comparator): After induction parturient in the ESPB underwent bilateral ESPB at the level of T7 using a linear ultrasound (US) transducer.
  Intravenous fentanyl patient control device 24-hour fentanyl consumption will be recorded.
  Interventions: Procedure: Erector Spinae Plane Block; Procedure: Intravenous fentanyl patient control device
- control group (Active Comparator): No regional anesthesia technique will be applied to the control group.
  Intravenous fentanyl patient control device 24-hour fentanyl consumption will be recorded.
  Interventions: Procedure: Intravenous fentanyl patient control device

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — The transducer was placed vertically 3cm lateral to the midline to visualize the muscles of the back, transverse process and the pleura in between the two transverse processes. After local infiltration of the needle insertion site with 2-3 ml of 2% lidocaine needle was inserted in cranial-caudal direction towards the transvers process using in plane technique until the needle cross all the muscles then interfascial injection of 20ml local anesthetics is done after ensuring negative aspiration, the procedure was repeated following the same steps on the other side of the back.
  Arms: ESP( Erector Spinae Plane Block)
Procedure: Intravenous fentanyl patient control device — 24-hour fentanyl consumption will be recorded.

SUMMARY:
The goal of this study is to evaluate the effect of ultrasound guided erector spinae plane block on postoperative pain and quality of recovery after laparoscopic colon surgery.

DETAILED DESCRIPTION:
.The goal of this study is to evaluate the effect of ultrasound guided erector spinae plane block on postoperative pain and quality of recovery after laparoscopic colon surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 70 years, with an American Society of Anesthesiologists physical status of 1 or 2, who were scheduled for laparoscopic colorectal operation

Exclusion Criteria:

* sensitivity to local anesthetic, bleeding disorders , receiving anticoagulant, body mass index (BMI) over 35/kg/m2 spine or chest wall deformity pregnancy tolerance to opioid analgesics inability to use patient-controlled analgesia (PCA)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
numerical rating scale on rest and cough | 24 hours after surgery
  In the recovery room, post op 6hours, post op 24 hours

SECONDARY OUTCOMES:
opioid consumption | 24 hours after surgery
  In the recovery room, post op 6hours, post op 24 hours
Quality of Recovery | 1day before operation, post op 24 hours
  pre operative QoR 40 scores compares
need for analgesics | 24 hours after surgery
  Number of patients who required analgesic in the first 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: hyunjeong kwack, md,phd, Study Director — Gachon University Gil Medical Center
Locations (1):
- Gachon University College of Medicine, Gil Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No